CLINICAL TRIAL: NCT03108443
Title: Novel Markers for Detecting Early Progression of Glaucoma
Status: Active, not recruiting | Type: Observational
Sponsor: Balwantray Chauhan (Other)
Responsible Party: Sponsor-Investigator, Balwantray Chauhan, Mathers Professor and Research Director, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: 1022071
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Glaucoma: Subjects identified as having glaucoma. No interventions will be performed.
  Interventions: Diagnostic Test: Optical Coherence tomography angiography
- Healthy controls: Subjects identified as having healthy eyes with no disease.
  Interventions: Diagnostic Test: Optical Coherence tomography angiography

INTERVENTIONS:
Diagnostic Test: Optical Coherence tomography angiography — All subjects will have OCT angiography imaging performed

SUMMARY:
Current methods of detecting glaucoma and monitoring its progression over time involve visual assessment of the optic nerve, thickness measurements of nerve tissue in the eye (using optical coherence tomography, OCT) as well as functional tests which measure peripheral, or side, vision. The objective of this study is to determine if a new technique of measuring blood flow in the eye, using OCT, can be used to better detect and/or monitor changes in glaucoma patients and suspects than these methods.

DETAILED DESCRIPTION:
Changes in the superficial optic nerve head (ONH) surface and loss of retinal nerve fibre layer (RNFL) thickness detected with clinical imaging are predictive of future visual field loss. Imaging of the deep ONH, the likely origin of glaucomatous damage, represents the next logical next step, but has eluded clinicians because of the lack of capable technology.

New advances in optical coherence tomography (OCT) imaging now offer an exciting opportunity to close the gap between the histomorphometric knowledge on deep ONH changes gained with research in experimental monkey glaucoma and imaging in clinical glaucoma.

There is compelling evidence that gross ONH and retinal hemodynamic changes are functional indicators of glaucoma progression. Accurate tracking of blood flow in the ONH is a logical step, but has evaded researchers for several reasons including the highly reflective ONH tissue which variably inhibits signal penetration making the complex nature of retinal and posterior ciliary contributions to ONH flow difficult to segregate. Even though glaucoma damage originates in the ONH, retinal ganglion cell (RGC) axons may show the earliest functional alterations as they have high metabolic demand and vulnerability to damage. Therefore, tracking blood flow in the RNFL, which is highly segmental and resolvable, could be a better and more sensitive approach compared to that in the ONH. The macula contains almost 50% of the entire RGC population; likewise, monitoring blood flow in the macular inner vascular plexus corresponding to the ganglion cell layer (GCL) is likely to be highly informative for glaucoma progression. OCT based angiography (OCTA), which maps vessel density in different retinal vascular beds with unparalleled axial resolution, will finally allow us to quantify highly localized parameters related to blood flow and identify patients with higher progression risk. Current data analysis of progression detection based on inter-subject or population-based variability models are inefficient, leading to false-positive and false-negative results. Innovative data analysis techniques that build accurate models of intra-subject variability will add cumulative value to the novel imaging markers for progression.

ELIGIBILITY:
Glaucoma Group

Inclusion Criteria:

* visual acuity ≥ 6/12
* glaucomatous ONH change
* glaucomatous visual field loss with a positive Glaucoma Hemifield Test

Exclusion Criteria:

* non-glaucomatous ocular disease
* chronic systemic disease or treatment affecting the visual field
* refraction exceeding 6 D equivalent sphere or 3 D astigmatism
* inability to provide informed consent

Control Group

Inclusion Criteria:

* visual acuity ≥ 6/12
* normal eye examination with intraocular pressure ≤ 21 mm Hg
* normal visual field and negative Glaucoma Hemifield Test

Exclusion Criteria:

* chronic ocular disease
* chronic systemic disease or treatment affecting the visual field
* refraction exceeding 6 D equivalent sphere or 3 D astigmatism
* inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Glaucoma patients recruited from a Primary Care Clinic Healthy control subjects recruited from the general population
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Blood flow | Changes over the 5 year course of the study
  Establish whether blood flow changes occur and if there are differences in the groups.

SECONDARY OUTCOMES:
Optic nerve head (ONH) anatomy | Changes over the 5 year course of the study
  Measure changes in the structure of the ONH

CONTACTS AND LOCATIONS:
Overall Officials: Balwantray Chauhan, PHD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Eye Care Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No